CLINICAL TRIAL: NCT07204470
Title: The Effects of Four Instant Maize Porridges on Satiety Measures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2410
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Satiety
Keywords: whole grain; appetite; glycemic index; leptin; ghrelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Whole grain maize porridge prepared with cold water (Experimental): White Star Whole Grain Instant Maize Porridge Original
  Interventions: Other: Breakfast cereal standardised to an isocaloric intake of approximately 350 kcal, consume entire portion within 15 minutes witnessed. No other food may be consumed during the 4 hour test period.
- Whole grain maize porridge prepared with hot water (Experimental): White Star Whole Grain Instant Maize Porridge Original
  Interventions: Other: Breakfast cereal standardised to an isocaloric intake of approximately 350 kcal, consume entire portion within 15 minutes witnessed. No other food may be consumed during the 4 hour test period.
- Smart Food (Experimental): FUTURELIFE Smart Food Original
  Interventions: Other: Breakfast cereal standardised to an isocaloric intake of approximately 350 kcal, consume entire portion within 15 minutes witnessed. No other food may be consumed during the 4 hour test period.
- Instant Maize Porridge - reduced sugar formulation (WSIP) (Experimental): White Star Instant Maize Porridge Original- reduced sugar formulation (WSIP)
  Interventions: Other: Breakfast cereal standardised to an isocaloric intake of approximately 350 kcal, consume entire portion within 15 minutes witnessed. No other food may be consumed during the 4 hour test period.

INTERVENTIONS:
Other: Breakfast cereal standardised to an isocaloric intake of approximately 350 kcal, consume entire portion within 15 minutes witnessed. No other food may be consumed during the 4 hour test period. — Cereal is in porridge form. One 350 ml bottle of water provided for the 4 hour test period 7:00-11:00 a.m.. Control dinner meal consumed the prior evening, then fast 10 hours overnight before visiting the test facility on four test days one week apart.

SUMMARY:
This study is designed to test the hypothesis that whole-grain forms of maize meal enhance and prolong satiety post-meal consumption.

ELIGIBILITY:
Inclusion Criteria:

* Availability to participate on the test days
* Interest and consent to participate in the study
* Participants must be willing to fast 10 hours overnight before the test breakfast meal (only water allowed)
* Products and meals high in fiber, alcohol and strenuous exercise should be avoided 24 hours before the test
* Age 18-35 years
* Healthy BMI: 18.5-24.9 kg/m2
* Equal split, males and females

Exclusion Criteria:

* Pregnancy; breast-feeding
* History of gastrointestinal disease having an impact on food absorption or digestion; anorexia nervosa or bulimia nervosa
* Anaemia
* Hypoglycaemia
* Cardiovascular disease; elevated plasma glucose; unstable thyroid function
* Abnormal/irregular menstrual cycle
* Substance abuse
* Being on medication which influences appetite
* Depression; smoking
* Participation in any weight altering program; weight gain or loss > 5 kg in 3 months prior to enrolment
* History of intestinal discomfort when consuming relatively small (e.g., <10g) amounts of non-digestible fibres
* Any known food allergies or intolerances such as wheat or soy; special diets prescribed by medical practitioner
* Any intensive physical training program

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Satiety -Appetite | On each of four testing days, in fasted state, immediately after the standardised breakfast (0), and at 120 and 240 min after the breakfast
  Self-reported appetite ratings using a 100 mm visual analog scale (VAS) questionnaire with 3 items: desire to eat rated from very weak to very strong, hunger rated from not at all to extremely, and fullness rated from not at all to extremely.
Satiety -Biomarkers: Leptin | On each of four test days at baseline following a 10 hour fast (Time 0), at 2 hours and 4 hours post ingestion of test porridge
  Blood by venipuncture to measure the appetite-regulating hormone leptin in nanograms per milliliter
Satiety -Biomarkers: Ghrelin | On each of four test days at baseline following a 10 hour fast (Time 0), at 2 hours and 4 hours post ingestion of test porridge
  Blood by venipuncture to measure the appetite-regulating hormone ghrelin in picograms per milliliter
Satiety - glycaemic parameters: Glucose | On each of four test days at baseline following a 10 hour fast (Time 0), at 2 hours and 4 hours post ingestion of test porridge
  Blood samples obtained by venipuncture in millimoles per liter
Satiety - glycaemic parameters: Insulin | On each of four test days at baseline following a 10 hour fast (Time 0), at 2 hours and 4 hours post ingestion of test porridge
  Serum samples obtained by venipuncture in microunits per milliliter

SECONDARY OUTCOMES:
Anthropometric measurements - BMI | Test Day 1 only prior to porridge consumption
  Body mass index calculated from kg weight and cm height
Anthropometric measurements - WHR | Test Day 1 only prior to porridge consumption
  Waist-hip ratio in centimeters
Anthropometric measurements - Fat Mass | Test Day 1 only prior to porridge consumption
  Body composition measurement
Dietary intake habits-QFFQ | The protocol allows for completion prior to the first test day, or instead at any one of the four test days. There is no particular time point requirement that it be done at baseline nor within a certain window after test meal consumption.
  Interviewer-administered, completed once using a quantified food frequency questionnaire (QFFQ) of 140 typically consumed food items by type/brand, cooking methods, frequency, and the amount of all food and drink consumed in the past 4 weeks converted to grams per week per food item
Dietary intake habits-24 hour recall | Completed at each of the four test days. There is no particular time point requirement that it be done at baseline nor within a certain window after test meal consumption.
  Using a quantified food frequency questionnaire (QFFQ)

CONTACTS AND LOCATIONS:
Overall Officials: Henrietta L de Kock, Principal Investigator — U Pretoria
Locations (1):
- U. Pretoria, Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: No